CLINICAL TRIAL: NCT02385773
Title: A Double Blind, Randomized, Placebo-Controlled Trial to Assess the Impact of the Nutritional Product PTM202 on Acute and Long-Term Recovery From Childhood Diarrheal Disease
Brief Title: Impact of the Nutritional Product PTM202 on Acute and Long-Term Recovery From Childhood Diarrheal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: PanTheryx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-1372
Record Dates: First submitted 2015-02-06; First posted 2015-03-11 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diarrhea
Keywords: colostrum; Immunoglobulin Y (IgY)
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTM202 (Experimental): PTM202
  Interventions: Dietary Supplement: PTM202
- Enfamil Puramino (Placebo Comparator): Formal Placebo
  Interventions: Dietary Supplement: Enfamil Puramino

INTERVENTIONS:
Dietary Supplement: PTM202 — Administration of study nutritional product once per day for 3 days starting immediately after enrollment
  Other Names: Conforta123
  Arms: PTM202
Dietary Supplement: Enfamil Puramino — Administration of 30 ml of Enfamil Puramino as placebo once per day for 3 days starting immediately after enrollment
  Arms: Enfamil Puramino

SUMMARY:
This trial will assess the impact of the nutritional product PTM202 on childhood diarrhea in Guatemalan children. The product is based on cow-milk colostrum and egg. The trial will enroll children between the ages of 6 months and 3 years and will assess the impact of the study nutrition product on the duration and severity of diarrhea and on weight recovery in the 4 weeks following the diarrheal episode. The investigators will be determining the etiology of the diarrhea episode to ascertain if the nutritional product works better for certain etiologies or has a non-specific benefit.

DETAILED DESCRIPTION:
This is a double-blind, randomized control trial of the nutritional product PTM202, which is a food product based on cow milk colostrum and eggs from hens that have been immunized against human diarrheal pathogens. Children between the ages of 6 months and 3 years will be enrolled at two sites in Guatemala who present with acute diarrhea. The study will have two strata according to the severity of the diarrhea.

The study product will be administered over 3 days, and the investigators will assess the impact on diarrhea duration and severity, and then follow subjects for 4 weeks to assess the impact of the nutritional product on weight gain following the episode, because poor weight gain is a major health problem in low-income countries. The investigators will also monitor for any adverse events during the trial.

The duration of participation will be 31 days for all subjects.

A stool sample will be collected at enrollment to ascertain the etiology of the diarrhea. A second sample will be collected at the end of the study to assess changes in pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent or legal guardian is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 6 months to 35 months.
* Presenting to care for acute diarrhea of 72 hours duration or less at the time of enrollment.
* Greater than 3 liquid stools in the previous 24 hours.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Additional inclusion for Arm 1: in addition to above, the subject will require or have already required > 8 hours of active rehydration in hospital or ER diarrheal ward, as determined by the attending physician.
* Additional inclusion for Arm 2: in addition to above, the subject will require or have already required < 8 hours of active rehydration in hospital or ER diarrheal ward, as determined by the attending physician.

Exclusion Criteria:

* Clinical condition for which oral intake of test product or placebo is contraindicated in opinion or attending physician.
* History of hypersensitivity or adverse reaction to milk or egg products.
* Condition improving in last 24 hours per parental report.
* Mild disease severity, defined as no recommended period of observed rehydration therapy per attending physician.
* Bloody Diarrhea at presentation.
* Severe malnutrition, defined as weight-for-age Z-score < -3 from median WHO published norms.
* Major congenital defects or serious chronic illness (neurologic, pulmonary, gastrointestinal liver, renal or endocrine).
* Receipt of probiotics in 72 hours prior to enrollment or recommended treatment with probiotics by attending physician
* Any confirmed or suspected immunosuppressive or immunodeficient condition including human immunodeficiency virus infection (HIV).
* Subject who, in the opinion of the investigator or sub-investigator, is unlikely to comply with the protocol, including capability to receive follow-up telephone calls or return for final visit.

Ages: 12 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 321 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea | Subjects will be followed for the duration of the diarrheal illness, with an expected average duration of 72 hours
  Duration in hours until subject has achieved a 12 hour period without diarrheal stools

SECONDARY OUTCOMES:
Weight gain after diarrhea | 2 weeks
  Weight will be assessed 14 days after the day 3 rehydrated baseline weight
Weight gain after diarrhea | 4 weeks
  Weight will be assessed 28 days after the day 3 rehydrated baseline weight

CONTACTS AND LOCATIONS:
Overall Officials: James T Gaensbauer, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- Guatemala (2):
  - Clínicas del Centro de Desarrollo Humano, Coatepeque
  - Hospital Roosevelt, Guatemala City

REFERENCES:
- [Derived] Gaensbauer JT, Melgar MA, Calvimontes DM, Lamb MM, Asturias EJ, Contreras-Roldan IL, Dominguez SR, Robinson CC, Berman S. Efficacy of a bovine colostrum and egg-based intervention in acute childhood diarrhoea in Guatemala: a randomised, double-blind, placebo-controlled trial. BMJ Glob Health. 2017 Dec 4;2(4):e000452. doi: 10.1136/bmjgh-2017-000452. eCollection 2017. PMID 29259822